CLINICAL TRIAL: NCT05190640
Title: Study to Evaluate the Efficacy of Asystems' Complete Calm Supplementation on Sleep Quality and Duration, Anxiety, and Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asystem, Inc. (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20221Asystem
Record Dates: First submitted 2021-12-31; First posted 2022-01-13 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Sleep; Stress; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): The dietary supplement (Asystems) is designed, and marketed commercially to be taken in servings of one gummy: one gummy a day for De-Stress Gummies and one gummy a day for Sleep Gummies.
  Interventions: Dietary Supplement: De-Stress Gummies

INTERVENTIONS:
Dietary Supplement: De-Stress Gummies — one gummy a day for De-Stress Gummies and one gummy a day for Sleep Gummies

SUMMARY:
This is an open-label observational single-arm clinical trial to study the efficacy of a commercial dietary supplement and its effect on sleep quality, sleep duration, anxiety, mood, and stress.

DETAILED DESCRIPTION:
It is hypothesized that the dietary supplement marketed as "Asystems Complete Calm" (consisting of De-Stress Gummies and Sleep Gummies) will improve subjective wellbeing in trial participants, through promoting restful sleep (looking at sleep quality and duration), and reducing stress and anxiety, while lifting up the participants' mood.

A total of 35 participants will be recruited for the trial following the screening. The trial will be fully remote, a technology platform will be utilized to screen, enroll and capture study data of the participants, and all participants will take the Complete Calm Product, consisting of the De-Stress Gummies (day) and Sleep Gummies (night) for four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male & Female between 24-45 years old
* Self-reported (undiagnosed) mild to moderate sleep issues
* Self-reported (undiagnosed) mild to moderate anxiety
* Self-reported stressful lifestyle
* Must be in good health (don't report any medical conditions asked in the screening questionnaire)
* Following a stable, consistent diet regimen
* Willing to maintain current dietary pattern, activity level, and stable body weight for the duration of the study, and refrain from any drastic lifestyle changes

Exclusion Criteria:

* Currently taking any prescription anti-depressants
* Currently receiving other psychotherapeutic treatment for anxiety or depression
* Severe chronic conditions including oncological conditions, psychiatric disease, or other
* Diagnosed insomnia
* Diagnosed anxiety or depression
* Food intolerances/allergies that require an epipen
* Females that are pregnant, want to become pregnant for the duration of the study, or who are breastfeeding

Ages: 24 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Change in sleep quality [Time Frame: Baseline to 4 weeks) | 4 weeks
  Survey-based assessment (0-5 scale with 0 being the lowest possible score and 5 being the highest) of changes in sleep quality between baseline and study intervention period.
Change in stress and anxiety [Time Frame: Baseline to 4 weeks) | 4 weeks
  Survey-based assessment (0-5 scale with 0 being the lowest possible score and 5 being the highest) of changes in stress/anxiety between baseline and study intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Mitschke, MSc, Principal Investigator — Citruslabs
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided